CLINICAL TRIAL: NCT00999401
Title: A Phase I Study of Oral Sapacitabine and Oral Seliciclib in Patients With Advanced Solid Tumors
Brief Title: A Study of Oral Sapacitabine and Oral Seliciclib in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC682-07
Record Dates: First submitted 2009-10-19; First posted 2009-10-21 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — sapacitabine; Roscovitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sapacitabine and seliciclib (Experimental): Sequential or concomitant administration of sapacitabine and seliciclib
  Interventions: Drug: sapacitabine and seliciclib

INTERVENTIONS:
Drug: sapacitabine and seliciclib — sequential or concomitant administration of sapacitabine and seliciclib
  Other Names: CYC682 and CYC202

SUMMARY:
A study of sequential administration of oral sapacitabine and oral Seliciclib in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the maximum tolerated dose (MTD) or recommended phase II doses of sapacitabine and seliciclib administered sequentially or concomitantly. The secondary objectives are to evaluate antitumor activity of this sequential or concomitant treatment and to explore the pharmacodynamic effect of this treatment in skin and peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* Incurable advanced solid tumors that are no longer responding to conventional therapy or for which no effective therapy exists; at the RD of Part 1, an extension cohort up to 20 patients with metastatic breast cancer who are known to be BRCA mutation carriers will be enrolled.
* Age 18 years or older
* ECOG 0-2
* Life expectancy ≥ 3 months
* Evaluable disease
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function
* At least 3 weeks from prior systemic treatments including investigational anti-cancer therapy, radiation therapy; and have recovered from prior toxicities
* Able to swallow capsules
* At least 3 weeks from major surgery
* Agree to practice effective contraception
* Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Previously untreated CNS metastases or progressive CNS metastases
* Currently receiving radiotherapy, biological therapy, or any other investigational agents
* Uncontrolled intercurrent illness including
* Pregnant or lactating women
* Known to be HIV-positive
* A history of active hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-04; Primary Completion 2019-07-16 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 1-3 months
  MTD of both sapacitabine and seliciclib administered sequentially in advanced solid tumor patients

SECONDARY OUTCOMES:
tumor response rate | 1-3 months
  Anti-tumor activity of the sequential treatment of sapacitabine and seliciclib in patients with advanced solid tumors.
pharmacodynamic effects in skin and peripheral mononuclear cells | 1-3 months
  PD effect of the sequential treatment of sapacitabine and seliciclib in patients with advanced solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, M.D., Principal Investigator — Dana-Farber Cancer Institute; Sara Tolaney, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Shapiro GI, et al. Responses to sequential sapacitabine and seliciclib in patients with BRCA-deficient solid tumors. Cancer Res April 15, 2013 73; LB-202.